CLINICAL TRIAL: NCT04552743
Title: Phase II Study of MGTA-145 in Combination With Plerixafor in the Mobilization of Hematopoietic Stem Cells for Autologous Transplantation in Patients With Multiple Myeloma
Brief Title: MGTA-145 + Plerixafor in the Mobilization of Hematopoietic Stem Cells for Autologous Transplantation in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Surbhi Sidana, MD (Other)
Responsible Party: Sponsor-Investigator, Surbhi Sidana, MD, Assistant Professor of Medicine (Blood and Marrow Transplantation and Cellular Therapy), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-57056; BMT362 (Other: OnCore)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Chemokine CXCL2; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MGTA-145 and Plerixafor HSC Mobilization (Experimental): Patients after screening will undergo baseline evaluation during the premobilization phase up to 30 days before mobilization. Patients will undergo sequential administration of plerixafor 0.24 mg/kg subcutaneously followed 2 hours later by MGTA-145 at 0.03 mg/kg intravenously (3 to10 minute infusion). This will be followed by apheresis. A second day of mobilization and apheresis will be pursued in patients who have not collected 6.0 x 106 CD34+ cells/kg in one session.
  Interventions: Drug: MGTA-145; Drug: Plerixafor

INTERVENTIONS:
Drug: MGTA-145 — A chemokine receptor type 2 (CXCR2) agonist protein, administered via intravenous (IV) infusion over 3 to 10 minutes.
  Other Names: GRO beta
Drug: Plerixafor — An azamacrocycle CXCR4 chemokine receptor antagonist, administered at 0.24 mg/kg subcutaneously, reduced to 0.16 mg/kg in patients with renal dysfunction (per package insert).
  Other Names: Mozobil; AMD 3100; LM-3100

SUMMARY:
This study evaluates a new drug MGTA-145 in combination with plerixafor (Mozobil) to mobilize stem cells into the peripheral blood for collection by apheresis. The stem cells will be used for autologous stem cell transplant for treatment of multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

1. To assess the efficacy of MGTA-145 in combination with plerixafor in mobilizing adequate number of hematopoietic stem cells (> 2 x 10e6 CD34+ cells/kg) in patients with multiple myeloma (MM) in preparation for autologous stem cell transplantation (ASCT).

SECONDARY OBJECTIVES

1. To assess the efficacy of MGTA-145 and plerixafor in mobilizing different Hematopoietic stem cells (HSCs) target goals in patients with MM in preparation for ASCT.
2. To assess the safety and tolerability of MGTA-145 and plerixafor for mobilizing HSCs in patients with MM.
3. To assess the engraftment rate and time to engraftment following ASCT after HSC mobilization with MGTA-145 and plerixafor in patients with MM undergoing upfront ASCT.
4. To assess rate of ongoing engraftment at Day 30 and 100 after stem cell infusion in patients with MM who are mobilized with MGTA-145 and plerixafor undergoing upfront ASCT.
5. To assess transplant and disease-related outcomes after mobilization of HSCs with MGTA-145 and plerixafor in patients with MM undergoing upfront ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (MM) per the International Myeloma Working Group (IMWG) criteria
* Eligible for autologous stem cell transplantation (ASCT) per institutional guidelines
* Within 1 year of start of therapy for multiple myeloma
* Cardiac and pulmonary status sufficient to undergo apheresis and transplantation per institutional transplant guidelines
* Calculated creatinine clearance > 30 mL/min, according to the Modification of Diet in Renal Disease (MDRD) formula.
* Absolute neutrophil count (ANC) > 1500 x 10e6/L
* Platelet count > 100,000 x 10e6/L
* Ability to understand and the willingness to sign a written informed consent document.
* Agreement to use an approved form of contraception for male patients or female patients of childbearing potential.

Exclusion Criteria:

* History of prior stem cell transplant for multiple myeloma or other indications
* Planned tandem stem cell transplant
* Prior history of failure to collect HSCs.
* Total bilirubin > 1.5x upper limit of normal (ULN) in the absence of a documented history of Gilbert's syndrome
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 3x ULN
* Known allergy to MGTA-145 or plerixafor.
* Lifetime exposure to lenalidomide or another immunomodulatory drug greater than 6 cumulative months of treatment, ie, > 6 cycles of 28 days or > 8cycles of 21 days
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Surbhi Sidana, MD, Principal Investigator — Stanford Medicine at Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sidana S, Bankova AK, Hosoya H, Kumar SK, Holmes TH, Tamaresis J, Le A, Muffly LS, Maysel-Auslender S, Johnston L, Arai S, Lowsky R, Meyer E, Rezvani A, Weng WK, Frank MJ, Shiraz P, Maecker HT, Lu Y, Miklos DB, Shizuru JA. Phase II study of novel CXCR2 agonist and Plerixafor for rapid stem cell mobilization in patients with multiple myeloma. Blood Cancer J. 2024 Oct 9;14(1):173. doi: 10.1038/s41408-024-01152-1. PMID 39384609

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 7
Age, Continuous [Median (Standard Deviation); unit: years] | 62.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants For Whom 2.0 x 10e6 CD34+ HSC Cells/kg Could be Collected in 1 or 2 Apheresis Harvests
Description: The study Primary Objective is to assess the efficacy of hematopoietic stem cells (HSC) mobilization with MGTA-145 in combination with plerixafor in patients with multiple myeloma (MM) in preparation for autologous stem cell transplantation (ASCT). The primary outcome was assessed as the number of participants for whom 2.0 x 10e6 CD34+ HSC cells/kg could be collected in 1 or 2 apheresis harvests, after mobilization with MGTA-145 and Plerixafor. The outcome is reported as the number of participants who achieved this level of HSC cells, a number without dispersion.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 25
Participants | 22

2. Secondary Outcome: Other Measures of Hematopoietic Stem Cell (HSC) Yield in the Apheresis Product
Description: The study Primary Objective is to assess the efficacy of hematopoietic stem cells (HSC) mobilization with MGTA-145 in combination with plerixafor in patients with multiple myeloma (MM) in preparation for autologous stem cell transplantation (ASCT). Other secondary outcomes were assessed as the number of participants for whom 2.0 or 4.0 x 10e6 CD34+ HSC cells/kg could be collected in the Day 1 apheresis harvest only, and for whom the total yield ≥ 4.0 or ≥ 6.0 x 106 CD34+ cells/kg. The outcome is reported as the number of participants who achieved these levels of HSC cells, a number without dispersion.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 25
Participants
  ≥ 2.0 x 10e6 CD34+ cells/kg on Day 1 | 17
  ≥ 4.0 x 10e6 CD34+ cells/kg on Day 1 | 9
  Total ≥ 4.0 x 10e6 CD34+ cells/kg | 17
  Total ≥ 6.0 x 10e6 CD34+ cells/kg | 10

3. Secondary Outcome: Time To Neutrophil Engraftment
Description: Neutrophil engraftment after hematopoietic stem cells (HSC) transplant (infusion) is an important measure of the medical benefit of the mobilization and hematopoietic stem cells (HSC) infusion procedure. Time to neutrophil engraftment is defined as the number of days from the day of stem cell infusion to the 1st day of 3 consecutive days that absolute neutrophil count (ANC) is ≥ 0.5 x 10e9/L. Only the participants that proceeded to the HSC infusion are included in this outcome, with the outcome is expressed as the median number of days with full range.
Time Frame: 15 days
Measure: Median (Full Range); unit: days
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 25
days | 12 [11 to 15]

4. Secondary Outcome: Maintenance of Neutrophil Engraftment [Absolute Neutrophil Count (ANC) ≥ 0.5 x 10e9/L]
Description: Maintenance of successful engraftment after initial engraftment is an important assessment of the value of the mobilization and hematopoietic stem cells (HSC) infusion procedure. For participants with successful neutrophil engraftment [absolute neutrophil count (ANC) ≥ 0.5 x 10e9/L], the outcome is reported as the number of participants that had maintained successful graft status [absolute neutrophil count (ANC) ≥ 0.5 x 10e9/L] at 30 days and 100 days after the infusion. The outcome is a number without dispersion.
Time Frame: 100 days
Population: This outcome is limited to participants that proceeded to the hematopoietic stem cell (HSC) infusion procedure, and with successful neutrophil engraftment.
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 19
Participants
  ANC ≥ 0.5 x 10e9/L at 30 days | 19
  ANC ≥ 0.5 x 10e9/L at 100 days | 19

5. Secondary Outcome: Time To Platelet Engraftment ≥ 20 x 10e9/L
Description: Platelet engraftment after hematopoietic stem cells (HSC) transplant (infusion) is an important measure of the medical benefit of the mobilization and hematopoietic stem cells (HSC) infusion procedure. Time to platelet engraftment ≥ 20 x 10e9/L is defined as the 1st day of 2 consecutive days that platelet count is ≥ 20 x 10e9/L, without transfusion in the prior 7 days. Only the participants that proceeded to the HSC infusion are included in this outcome, with the outcome is expressed as the median number of days with full range.
Time Frame: 33 days
Population: This outcome is limited to participants that proceeded to the hematopoietic stem cell (HSC) infusion procedure.
Measure: Median (Full Range); unit: days
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 19
days | 18 [15 to 33]

6. Secondary Outcome: Time To Platelet Engraftment ≥ 50 x 10e9/L
Description: Platelet engraftment after hematopoietic stem cells (HSC) transplant (infusion) is an important measure of the medical benefit of the mobilization and hematopoietic stem cells (HSC) infusion procedure. Time to platelet engraftment ≥ 50 x 10e9/L s defined as the 1st day that platelet count is ≥ 50 x 10e9/L, without transfusion in the prior 48 hours. Only the participants that proceeded to the HSC infusion are included in this outcome, with the outcome is expressed as the median number of days, with full range.
Time Frame: 44 days
Population: This outcome is limited to participants that proceeded to the hematopoietic stem cell (HSC) infusion procedure.
Measure: Median (Full Range); unit: days
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 19
days | 20 [13 to 34]

7. Secondary Outcome: Infusion-related Toxicities
Description: Infusion-related toxicities are adverse events considered at least possibly-related to the study treatments MGTA-145, assessed from Baseline to 7 days after mobilization. The outcome is reported as a listing of the preferred terms for the "at least possibly-related" adverse events, with outcome being the number of adverse events of that preferred term. The outcome is a listing of numbers without dispersion.
Time Frame: 7 days after mobilization procedure
Measure: Number; unit: adverse events
Groups:
- Number of Events: Number of adverse events by preferred term experienced by participants receiving MGTA-145 and Plerixafor
Arm/Group | Number of Events
Number analyzed (Participants) | 25
adverse events
  Pain | 11
  Aspartate/alanine aminotransferase increase | 1
  Nausea | 2
  Headache | 1
  Hyperhidrosis | 1
  Low platelet count | 2
  Vomiting | 1
  Poor Graft Function (beyond 7 days post-mobilization) | 1

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is an important assessment of the value of the mobilization and hematopoietic stem cells (HSC) infusion procedure. For participants that received the HSC infusion, the outcome is reported as the number of participants who remained alive and were without tumor progression, at 100 days after the infusion. The outcome is a number without dispersion.
Time Frame: 100 days after infusion procedure
Population: This outcome is limited to participants that proceeded to the hematopoietic stem cell (HSC) infusion procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 19
Participants | 18

9. Secondary Outcome: Transplant-related Mortality
Description: Transplant-related mortality is an important assessment of the value of the mobilization and hematopoietic stem cells (HSC) infusion procedure. For participants that received the HSC infusion, the outcome is reported as the number of participants who had expired for any reason considered at least possibly related to the transplant / infusion procedure, within 100 days of the infusion. The outcome is a number without dispersion.
Time Frame: 100 days after infusion procedure
Population: This outcome is limited to participants that proceeded to the hematopoietic stem cell (HSC) infusion procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 19
Participants | 0

10. Secondary Outcome: Non-relapse-related Mortality
Description: For participants that received the HSC infusion, the outcome is reported as the number of participants who had expired for any reason except disease relapse/progression, within 100 days of the infusion. The outcome is a number without dispersion.
Time Frame: 100 days after infusion procedure
Population: This outcome is limited to participants that proceeded to the hematopoietic stem cell (HSC) infusion procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 19
Participants | 0

11. Secondary Outcome: Overall Survival (OS)
Description: Only patients proceeding with upfront transplant will be assessed. Overall survival is defined as duration from start of the ASCT to death (regardless of cause of death). This will be assessed from start of transplant and OS rates will be reported at day100 following transplant in patients undergoing upfront transplant.
  Overall survival (OS) is an important assessment of the value of the mobilization and hematopoietic stem cells (HSC) infusion procedure. For participants that received the HSC infusion, the outcome is reported as the number of participants who remained alive at 100 days after the infusion. The outcome is a number without dispersion.
Time Frame: 100 days after infusion procedure
Population: This outcome is limited to participants that proceeded to the hematopoietic stem cell (HSC) infusion procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Time Frame: Per protocol at 7.2.3, adverse events were collected from baseline through 30 days after the last dose of MGTA-145, up to 32 days.
Arm/Group | MGTA-145 and Plerixafor HSC Mobilization
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 25/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MGTA-145 and Plerixafor HSC Mobilization (N=25)
Pain (General disorders) | 13 (16)
Fatigue (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Other - Poor Graft Function (anemia, neutropenia, thrombocytopenia) (Blood and lymphatic system disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 7 (8)
Dizziness (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT04552743/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04552743/ICF_001.pdf